CLINICAL TRIAL: NCT00743158
Title: Transfer Impedance in Cystic Fibrosis (Ztr)
Brief Title: Transfer Impedance in Cystic Fibrosis
Acronym: Ztr
Status: Withdrawn | Type: Observational
Why Stopped: PI determination
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Thomas Martin, Assistant Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: X08-01-0060
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Cystic Fibrosis
Keywords: ztr; transfer impedance; cystic fibrosis; pulmonary function test; pft
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
This study aims to determine whether respiratory system transfer impedance (Ztr) may fill an important clinical function by providing a reproducible, valid, and sensitive measure of airway obstruction in people with CF.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 2 to 25 Confirmed diagnosis of Cystic Fibrosis

Exclusion Criteria:

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cystic Fibrosis Patients
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2011-03-03 (Actual); Study Completion 2011-03-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens Hospital, Boston, Boston, Massachusetts, United States